CLINICAL TRIAL: NCT03626701
Title: A Prospective Multicenter Randomized Controlled Clinical Study to Investigate the Safety and Effectiveness of RES® (Regenerative Epidermal Suspension) Prepared With the RECELL® Device Compared to Standard of Care Dressings for Treatment of Partial-thickness Burns in Infants, Children and Adolescents (Aged 1-16 Years)
Brief Title: RES® Prepared With RECELL® Compared to Standard of Care Dressings of Partial-thickness Burns in Ages 1-16 Years
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: In June 2021, the US FDA approved expanded use of the RECELL System for treatment of acute full-thickness thermal burns in patients 1-month of age and older (removing the prior limitation of use in patients younger than 18 years of age).
Sponsor: Avita Medical (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CTP006-2; RESTORE KIDS (Other: AVITA Medical)
Record Dates: First submitted 2018-07-20; First posted 2018-08-13 (Actual); Results first posted 2023-06-26 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Burns
Keywords: Pediatric; Burns; Partial-thickness
MeSH Terms: conditions — Burns

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: 1. Blinded Evaluator/Observer - local burn specialist
  2. Independent Reviewer
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- RECELL® Autologous Cell Harvesting Device (Experimental): RECELL + Telfa™ Clear and Xeroform™ dressings
  Conventional autografting (only when indicated)
  Interventions: Device: RES (Regenerative Epidermal Suspension) prepared using the RECELL® Autologous Cell Harvesting Device; Procedure: Conventional autografting (only when indicated)
- Mepilex® Ag Wound Dressing (Active Comparator): Mepilex® Ag Wound Dressing
  Conventional autografting (only when indicated)
  Interventions: Combination Product: Mepilex® Ag Wound Dressing; Procedure: Conventional autografting (only when indicated)

INTERVENTIONS:
Device: RES (Regenerative Epidermal Suspension) prepared using the RECELL® Autologous Cell Harvesting Device — Application of RES prepared using the RECELL® Autologous Cell Harvesting Device along with Telfa™ Clear primary and Xeroform™ secondary wound dressings.
  Arms: RECELL® Autologous Cell Harvesting Device
Combination Product: Mepilex® Ag Wound Dressing — Application of Mepilex® Ag Wound Dressing
  Arms: Mepilex® Ag Wound Dressing
Procedure: Conventional autografting (only when indicated) — When indicated, conventional autografting in accordance with Investigator's standard practice

SUMMARY:
A prospective, parallel-arm, randomized (1:1) multicenter trial to demonstrate that RECELL treatment of partial-thickness burn injuries, can safely and effectively increase the incidence of Day 10 healing compared with a standardized wound dressing.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 1 through 16 years (inclusive) with a partial-thickness thermal burn injury.
2. The patient has a thermal burn injury that is:

   1. ≤ 30% TBSA (exclusive of superficial areas) and
   2. ≤ 10% of the burn injury TBSA is a full-thickness burn.
3. The Index Burn must be a clean partial-thickness burn injury > or = to 160 cm2 and between 2-20% BSA (inclusive).
4. The Index Burn may not cover the face, hand, foot or perineum/genitalia (Note: a patient with wounds in these areas may be enrolled but the Index Burn Area may not include these areas).
5. The patient and/or guardian agrees to comply with all compulsory study procedures and visit schedule.
6. The patient and/or parent/guardian agrees to abstain from any other treatment for closure of the Index Burn for the duration of the study, unless medically necessary.
7. The patient and/or parent/guardian agrees to abstain from enrollment in any other interventional clinical trial for the duration of the study.
8. In the opinion of the investigator, the patient and/or parent/guardian must be able to:

   1. Understand the full nature and purpose of the study, including possible risks and adverse events,
   2. Understand instruction, and
   3. Provide voluntary informed written consent/assent as appropriate for study participation.

Exclusion Criteria:

1. Not able to understand English or Spanish.
2. Burns caused by chemicals, electricity or radiation.
3. Patients presenting with only 3rd-degree/full-thickness wounds which require immediate autografting.
4. Burn injury has had prior treatment for definitive closure.
5. Patients for whom use of sedation/general anesthesia is not medically appropriate.
6. Superficial/trivial burns or burns that in the investigator's opinion appear to be healing sufficiently such that care under this protocol would be inappropriate.
7. Patient requires immediate or staged surgical procedures for closure of their partial-thickness burns.
8. Conditions, e.g., previous burn injury to study area, poor nutritional status, poorly controlled diabetes mellitus (HbA1c >9%), that in the investigator's opinion may compromise subject safety or trial objectives.
9. Current use of medications, e.g., immunosuppressive agents (excluding inhaled corticosteroids), that in the investigator's opinion may compromise subject safety or trial objectives.
10. Inhalation injury.
11. Active infection, cellulitis or need for immediate grafting at the planned treatment areas.
12. Concerns for parent/guardian's ability to provide appropriate follow-up care.
13. Subjects with a known hypersensitivity to trypsin or compound sodium lactate for irrigation solution.
14. Subjects with a known sensitivity to silver.
15. In post-pubescent girls, pregnant or breast-feeding (pregnancy test should be performed in accordance with local institutional requirements).
16. Immediate life-threatening condition or life expectancy less than one year.
17. Previous randomization within this investigation.

Post-Randomization Inclusion Criteria (prior to treatment):

1. Patient randomized (and will be treated) within 72 hours from the time of the burn injury.
2. Patient continues to meet all pre-randomization inclusion criteria.

Post-Randomization Exclusion Criteria (prior to treatment):

1. Incidental finding of any pre-randomization exclusion criteria.

Consented subjects who do not meet the post-randomization eligibility criteria and did not receive study treatment will be followed through the Day 28 visit and then withdrawn from the study. The criteria for which exclusion was based will be documented.

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2021-06-23 (Actual); Study Completion 2022-06-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Arizona Burn Center / Valleywise Health, Phoenix, Arizona
  - University of South Florida Tampa General Hospital, Tampa, Florida
  - University Medical Center New Orleans, New Orleans, Louisiana
  - University of North Carolina, Chapel Hill, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Evan Hayes Burn Center, Virginia Commonwealth University, Richmond, Virginia
  - University of Washington Regional Burn Center at Harborview Medical Center, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- RECELL® Autologous Cell Harvesting Device: RECELL + Telfa™ Clear and Xeroform™ dressings
  Conventional autografting (only when indicated)
  RES (Regenerative Epidermal Suspension) prepared using the RECELL® Autologous Cell Harvesting Device: Application of RES prepared using the RECELL® Autologous Cell Harvesting Device along with Telfa™ Clear primary and Xeroform™ secondary wound dressings.
  Conventional autografting (only when indicated): When indicated, conventional autografting in accordance with Investigator's standard practice
- Mepilex® Ag Wound Dressing: Mepilex® Ag Wound Dressing
  Conventional autografting (only when indicated)
  Mepilex® Ag Wound Dressing: Application of Mepilex® Ag Wound Dressing
  Conventional autografting (only when indicated): When indicated, conventional autografting in accordance with Investigator's standard practice
Period: Overall Study
Arm/Group | RECELL® Autologous Cell Harvesting Device | Mepilex® Ag Wound Dressing
Started | 13 | 6
Completed | 9 | 5
Not Completed | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RECELL® Autologous Cell Harvesting Device | Mepilex® Ag Wound Dressing | Total
Number analyzed (Participants) | 13 | 6 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.0 (5.92) | 6.5 (3.78) | 8.9 (5.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 10 | 3 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 12 | 6 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 3 | 8
  White | 6 | 1 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 13 | 6 | 19

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Index Burns With Day 10 Healing
Description: Day 10 healing will be evaluated by an observer blinded to treatment allocation with confirmation at Day 28
Time Frame: 10 Days post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | RECELL® Autologous Cell Harvesting Device | Mepilex® Ag Wound Dressing
Number analyzed (Participants) | 13 | 5
Participants | 6 | 2

2. Secondary Outcome: Incidence of Day 21 Healing of the Index Burn
Description: Incidence of Day 21 healing of the Index Burn confirmed on Day 28
Time Frame: Day 21, confirmed on Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | RECELL® Autologous Cell Harvesting Device | Mepilex® Ag Wound Dressing
Number analyzed (Participants) | 12 | 4
Participants | 7 | 2

3. Secondary Outcome: Incidence of Conventional Autografting to Achieve Healing of the Index Burn
Description: Incidence of conventional autografting to achieve healing of the Index Burn
Time Frame: Through Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | RECELL® Autologous Cell Harvesting Device | Mepilex® Ag Wound Dressing
Number analyzed (Participants) | 13 | 6
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | RECELL® Autologous Cell Harvesting Device | Mepilex® Ag Wound Dressing
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/13 | 1/6
Other Adverse Events (participants affected / at risk) | 6/13 | 3/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RECELL® Autologous Cell Harvesting Device (N=13) | Mepilex® Ag Wound Dressing (N=6)
Impaired Healing (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RECELL® Autologous Cell Harvesting Device (N=13) | Mepilex® Ag Wound Dressing (N=6)
Impaired Healing (General disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
Community Acquired Infection (Infections and infestations) | 1 (1) | 0 (0)
Skin Infection (Infections and infestations) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypertrophic Scar (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-11): https://cdn.clinicaltrials.gov/large-docs/01/NCT03626701/Prot_SAP_002.pdf